CLINICAL TRIAL: NCT00432185
Title: An Open-label, Multi-center, Dose-escalation, Cohort Study to Determine the Maximum Tolerated Dose and Safety of PEP005 Topical Gel Given as Either a Single Application (on Day 1) or as Two Applications (on Day 1 and Day 8) to a Superficial Basal Cell Carcinoma (sBCC) on the Trunk.
Brief Title: To Determine the Maximum Tolerated Dose Level (MTD) of PEP005 Topical Gel in Patients With sBCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-009
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Superficial Basal Cell Carcinoma
Keywords: sBCC; Topical; Dermatology
MeSH Terms: interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): One day treatment
  Interventions: Drug: PEP005
- 2 (Active Comparator): Two day treatment
  Interventions: Drug: PEP005

INTERVENTIONS:
Drug: PEP005 — 0.25% PEP005 Gel

SUMMARY:
The purpose of this study is to determine maximum tolerated dose level (MTD) of PEP005 Topical Gel for the treatment of superficial basal cell carcinoma on the trunk

DETAILED DESCRIPTION:
Basal cell carcinomas (BCCs) are a common skin problem largely caused by long term sun exposure. Current treatments include surgery, curettage/desiccation and simple excision, which are often cosmetically disfiguring. Non-invasive alternative therapy for treatment of BCC lesions is thus being researched. Sap from the plant Euphorbia peplus has been used for many years in Australia as a "folk" remedy to treat a number of skin conditions. The active component of Euphorbia peplus has been isolated and made into a gel applied directly to the skin by Peplin Opeation Pty Ltd.

The proposed study follows a previously conducted 12 week study in sBCC, PEP005-003. This was a two dose schedule evaluating doses up to 0.05%. Histological clearance rate at the end of study was 71% for the 0.05% concentration on the Day 1, Day 2 schedule compared with 0% in the vehicle group.

The proposed study aims to determine the maximum tolerated dose level (MTD) of PEP005 Topical Gel, in patients, when administered either as a single application or as two applications to a selected superficial basal cell carcinoma lesion with a 3 month follow up.

ELIGIBILITY:
1. Male or female patients at least 18 years of age.
2. A primary clinically diagnosed and histologically confirmed sBCC lesion located on the trunk which is suitable for excision the histological diagnosis should be made no more than 60 days prior to the screening visit the biopsy specimen should have removed no more that 20% of the total tumour mass
3. Ability to follow study instructions and likely to complete all study requirements.
4. Written informed consent has been obtained.
5. Agreement from the patient to allow photographs of the selected lesion to be taken and used as part of the study data package.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose level (MTD) through incidence of treatment related AEs, local skin reactions and pigmentation and scarring. | 85 days

SECONDARY OUTCOMES:
Efficacy (complete sBCC clearance rate and composite sBCC clearance rate) | 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, Study Director — Peplin
Locations (9):
- United States (9):
  - Alta Dermatology, Mesa, Arizona
  - Dermatology Specialists Inc., Oceanside, California
  - Skin Surgery Medical Group Inc., San Diego, California
  - Colorado Medical Research Center, Denver, Colorado
  - Advanced Dermatology and Cosmetic Surgery, Clermont, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Minnesota Clinical Studies Center, Fridley, Minnesota
  - Dermatology Associates of Rochester, Rochester, New York
  - Rivergate Dermatology and Skin Care Center, Goodlettsville, Tennessee

REFERENCES:
- [Result] Gross K. Safety and efficacy of ingenol mebutate (PEP005) gel for topical treatment of superficial basal cell carcinoma. J Am Acad Dermatol 2009; 60(3, Suppl. 1): AB141; P2928
- [Result] Gross K, Schmieder GJ, Tu J. Maximum Tolerated Dose and Safety of PEP005 (ingenol mebutate) Gel for Topical Treatment of Superficial Basal Cell Carcinoma. Summer Academy, American Academy of Dermatology meeting, Boston, MA, 2009. 2009: Poster no. 1902 (31 p.)
- See also: Central IRB — http://www.quorumreview.com